CLINICAL TRIAL: NCT02418728
Title: The Contribution of Atrial Natriuretic Peptide in Lipid Mobilization of Subjects With Obesity, Both During Rest and Exercise
Brief Title: The Role of Atrial Natriuretic Peptide in the Lipolytic Process: Effect of Obesity and Exercise
Acronym: BALO
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, prof. dr., Hasselt University
Other Study IDs: CME2014 /450
Record Dates: First submitted 2015-03-17; First posted 2015-04-16 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: obesity; adipose tissue lipolysis; lipolysis; microdialysis; atrial natriuretic peptide
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- persons with obesity
  Interventions: Other: subcutaneous adipose tissue microdialysis under local beta/alpha blockade
- lean persons
  Interventions: Other: subcutaneous adipose tissue microdialysis under local beta/alpha blockade

INTERVENTIONS:
Other: subcutaneous adipose tissue microdialysis under local beta/alpha blockade — adipose tissue lipolysis under local beta/alpha blockade in abdominal subcutaneous adipose tissue, using microdialysis

SUMMARY:
In the developing countries, obesity prevalence is on a dramatic rise. Obesity is related to co-morbidities and as a result, obesity significantly shortens life expectancy and lowers quality of life. To prevent this, participation in exercise or training programs is absolutely necessary, in order to generate adipose tissue mass loss. The amount of adipose tissue mass loss is, amongst others, dependent on lipolysis which is under endocrine regulation by, mainly, catecholamines, insulin and atrial natriuretic peptide. However, large variations in adipose tissue mass loss and gain are likely in obese subjects, possibly due to a decreased lipolytic effect of these hormones (as was shown for catecholamines in the subcutaneous adipose tissue of obese subjects). However, the relative contribution of atrial natriuretic peptide in the lipolytic process remains elusive, particularly in subjects with obesity, which show an increased plasma expression of atrial natriuretic peptide.

The aim of the present study is to observe the contribution of atrial natriuretic peptide in the subcutaneous adipose tissue of obese subjects. This will be tested by measurements of extracellular glycerol levels (by microdialysis) in the subcutaneous adipose tissue in situ at rest and during endurance exercise under local beta- and alpha-blockade.

Eventually, the knowledge gained from this research will contribute to the optimization of exercise programs for people with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obese group: BMI > 30 kg/m², sedentary (no regular physical activity last 6 months), insulin sensitive or insulin resistant
* Lean controls: BMI > 18.5 kg/m² and < 25 kg/m², regular physical activity, insulin sensitive

Exclusion Criteria:

* Regular glucose lowering medication or beta blockade medication
* Presence of chronical diseases
* Orthopedic or neurological problems

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: subjects with obesity
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Subcutaneous adipose tissue microdialysis | week 1
  abdominal subcutaneous adipose tissue microdialysis during rest and exercise; basal + under local alpha- and beta-blockade.
Atrial natriuretic peptide (ANP) Response | week 1
  measurement systemic ANP response (venous blood sampling)

SECONDARY OUTCOMES:
Central insulin sensitivity | screening
  Fasting serum insulin, homeostasis model assessment insulin resistance and measures of central insulin sensitivity derived from an oral glucose tolerance test (75g)
Echocardiography | Day 1
  heart function by means of standard echocardiography
Maximal oxygen uptake (ml/O2/kg/min) | Day 1
  measured using indirect calorimetry and an incremental bicycle protocol
Anthropometry | screening
  body composition, measured using dual x-ray absorptiometry, height, weight, waist and hip circumference
Abdominal subcutaneous adipose tissue biopsy | week 1
  biochemical, proteomics and morphological analyses

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Blaak, prof. dr., Principal Investigator — Maastricht University; Kenneth Verboven, drs, Study Chair — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Belgium

IPD SHARING:
Plan to Share IPD: Undecided